CLINICAL TRIAL: NCT02040519
Title: Time of Onset and Time of Offset of Sacral Neuromodulation Effect - "Wash in - Wash Out"
Brief Title: Time of Effect Onset in Treating Overactive Bladder or Non Obstructive Urinary Retention by Sacral Neuromodulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL44879.068.13
Record Dates: First submitted 2014-01-13; First posted 2014-01-20 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Overactive Bladder; Non Obstructive Urinary Retention
Keywords: Overactive bladder; Non obstructive urinary retention; Sacral neuromodulation
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Evaluation by voiding diaries (Experimental)
  Interventions: Behavioral: Filling out voiding diaries.

INTERVENTIONS:
Behavioral: Filling out voiding diaries.

SUMMARY:
Sacral neuromodulation (SNM) is a minimally invasive secondary treatment for overactive bladder syndrome (OAB) or for non-obstructive urinary retention (NOR), when refractory to conservative treatment. Success rates range from 70 to 80%, and good long-term results are reported. The working mechanism of SNM is not completely understood, and the only prognostic factor for good response to this treatment is a successful test stimulation period. There is no consensus on the duration of this test stimulation period. The experience in our clinic during test stimulation period is that for responders it takes up to one week to achieve maximal effect, after the system is turned 'on'. On the other hand the investigators notice that after turning the neuromodulation system 'off', it will take a few hours for symptoms to return to the baseline situation. The fact is: no information concerning the so called "time of onset" and "time of offset" (or popular called: wash-in / wash-out) of sacral neuromodulation is available in current literature.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in this study, a subject must meet all of the following criteria: Patients should have been diagnosed with overactive bladder syndrome and should be put on the waiting list for scheduling treatment with sacral neuromodulation.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* patients receiving neurological or psychiatric medication without being diagnosed with a neurological or psychiatric disease
* patients who have been treated by means of bladder wall botulin toxin injections in the previous year
* patients with evident subsequent complaints of bladder pain syndrome or other pelvic pain

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-02-06 (Actual); Study Completion 2017-02-06 (Actual)

PRIMARY OUTCOMES:
Time of onset of effect of treatment with sacral neuromodulation | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: G. A. van Koeveringe, urologist, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands